CLINICAL TRIAL: NCT00953667
Title: The Genetics of Evoked Responses to Niacin and Endotoxemia: The GENE Study
Acronym: GENE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 805670
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Endotoxins; Niacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Niacin and Endotoxin (Experimental): All subjects are expected to have the same interventions- Niacin and Endotoxin.
  Interventions: Drug: Immediate Release Niacin, Extended Release Niacin, Endotoxin

INTERVENTIONS:
Drug: Immediate Release Niacin, Extended Release Niacin, Endotoxin — Subjects receive a one-time 1000mg dose of immediate release Niacin (Niacor pills), a one-time 1000mg dose of extended release Niacin (Niaspan pill) and one-time 1ng/kg injection of endotoxin (LPS).
  Other Names: Niacor; Niaspan

SUMMARY:
The purpose of this study is to determine genetic factors that affect responses to niacin therapy and endotoxemia in healthy volunteers.

DETAILED DESCRIPTION:
Niacin is a vitamin that has beneficial effects on cholesterol (a type of fat in the blood) when used in high doses. Different people respond differently to cholesterol lowering doses of niacin, some people have a side effect termed flushing (similar to a hot flash) while others do not and some people have more pronounced effects on cholesterol. Endotoxin or lipopolysaccharide (LPS) is a small part of bacteria (that is no longer living) that can cause many of the effects similar to bacterial infections in humans. However, it can be administered in very small amounts to produce a mild inflammatory response much the same as a 'flu-like" illness. Within 1 ½ -3 hours after giving LPS by vein, a response consisting of fever, chills, headache, nausea and vomiting and generalized aches and pains will occur which lasts up to 6-8 hours. In addition to the flu like symptoms, the inflammation causes changes in cholesterol, triglycerides and glucose clearance. Different people respond differently to endotoxin and inflammation. We are performing this study to see if there are genetic factors that predict how people will respond to niacin and to endotoxin and its inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

1. Men and non-pregnant/lactating women between the ages of 18 and 45.
2. Self reported African American or Caucasian racial-ethnic background.
3. Body Mass Index (BMI) of ≥ 18 and ≤ 30.
4. Participants who are able to give written informed consent and willing to comply with all study-related procedures.

Exclusion Criteria:

1. Known clinically manifest atherosclerotic cardiovascular disease, including coronary disease, cerebrovascular disease, or peripheral vascular disease.
2. History of diabetes mellitus.
3. Fasting glucose > 126 mg/dL.
4. History of a non-skin malignancy within the previous 5 years.
5. Renal insufficiency as defined by creatinine > 1.5 mg/dl at Screening Visit.
6. History of liver disease or abnormal liver function tests (LFTs) (AST, ALT, Alk. Phos., GGT > 1.5x upper limit of normal (ULN); bilirubin > 2x ULN) at Screening Visit.
7. Men who are unwilling to limit alcohol consumption to <14 alcoholic drinks per week or < 4 alcoholic drinks per occasion (AMA / NIAAA criteria for "at risk" usage levels) while participating in the study.
8. Women who are unwilling to limit alcohol consumption to < 7 alcoholic drinks per week or < 3 alcoholic drinks per occasion (AMA / NIAAA criteria for "at risk" usage levels) while participating in the study.
9. Total white blood cell count less than or equal to 3.0 THO/uL.
10. Hemoglobin below 11.0 g/dL.
11. Any major active rheumatologic, pulmonary, or dermatologic disease or inflammatory condition or minor active infection.
12. History of HIV positive.
13. First degree family history of premature cardiovascular disease event (father or brother if diagnosed at before 55 years of age; mother or sister if diagnosed before 65 years of age).
14. Patients who have undergone any organ transplant.
15. Individuals who currently use tobacco products or have done so in the previous 30 days.
16. Treatment with aspirin, non-steroidal anti-inflammatory drugs (NSAIDs), COX-2 inhibitors, steroids or any immunomodulatory therapy 2 weeks prior to the Screening Visit.
17. Treatment with statins, fibrates or niacin 4 weeks prior to the Screening Visit.
18. Current daily use of Vitamin C > 1000 mg, Beta carotene > 1000 IU, vitamin A > 5000 IU, vitamin E > 400 IU, and selenium > 200 mcg.
19. Positive urine pregnancy at the Screening Visit.
20. Participation in another clinical trial within the previous 6 weeks prior to the Screening Visit.
21. Poorly controlled blood pressure (BP > 160/110) or on any anti-hypertensive medications.
22. A diagnosis of metabolic syndrome using updated 2004 NCEP ATPIII criteria.
23. A history of severe lactose intolerance (e.g., intolerance of any milk intake).
24. Any medical condition or abnormal laboratory value that is judged clinically significant by an investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2007-06; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muredach P Reilly, M.B., MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Ferguson JF, Xue C, Gao Y, Tian T, Shi J, Zhang X, Wang Y, Li YD, Wei Z, Li M, Zhang H, Reilly MP. Tissue-Specific Differential Expression of Novel Genes and Long Intergenic Noncoding RNAs in Humans With Extreme Response to Evoked Endotoxemia. Circ Genom Precis Med. 2018 Nov;11(11):e001907. doi: 10.1161/CIRCGEN.117.001907. PMID 30571184
- [Derived] Ferguson JF, Shah RY, Shah R, Mehta NN, Rickels MR, Reilly MP. Activation of innate immunity modulates insulin sensitivity, glucose effectiveness and pancreatic beta-cell function in both African ancestry and European ancestry healthy humans. Metabolism. 2015 Apr;64(4):513-520. doi: 10.1016/j.metabol.2014.12.007. Epub 2014 Dec 26. PMID 25579865
- [Derived] Ferguson JF, Ryan MF, Gibney ER, Brennan L, Roche HM, Reilly MP. Dietary isoflavone intake is associated with evoked responses to inflammatory cardiometabolic stimuli and improved glucose homeostasis in healthy volunteers. Nutr Metab Cardiovasc Dis. 2014 Sep;24(9):996-1003. doi: 10.1016/j.numecd.2014.03.010. Epub 2014 Apr 18. PMID 24875672
- [Derived] Liu Y, Ferguson JF, Xue C, Ballantyne RL, Silverman IM, Gosai SJ, Serfecz J, Morley MP, Gregory BD, Li M, Reilly MP. Tissue-specific RNA-Seq in human evoked inflammation identifies blood and adipose LincRNA signatures of cardiometabolic diseases. Arterioscler Thromb Vasc Biol. 2014 Apr;34(4):902-12. doi: 10.1161/ATVBAHA.113.303123. Epub 2014 Feb 6. PMID 24504737
- [Derived] Ferguson JF, Patel PN, Shah RY, Mulvey CK, Gadi R, Nijjar PS, Usman HM, Mehta NN, Shah R, Master SR, Propert KJ, Reilly MP. Race and gender variation in response to evoked inflammation. J Transl Med. 2013 Mar 12;11:63. doi: 10.1186/1479-5876-11-63. PMID 23497455

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 400 subjects were enrolled over an approximate 3.5 year period in order to reach target of about 300 subjects completing all visits. Study ended with 277 subjects completing all visits.
Pre-assignment Details: All subjects received niacin and LPS doses. There were no separate arms.
Period: Overall Study
Arm/Group | Niacin and Endotoxin
Started | 400
Completed | 277
Not Completed | 123
Not completed — Lost to Follow-up | 11
Not completed — Physician Decision | 35
Not completed — Withdrawal by Subject | 63
Not completed — Adverse Event | 10
Not completed — poor venous access,unable to draw blood | 4

BASELINE CHARACTERISTICS:
Arm/Group | Niacin and Endotoxin
Number analyzed (Participants) | 400
Age, Continuous [Mean (Full Range); unit: years] | 25.42 [18 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 198
  Male | 202
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 143
  White | 255
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Baseline and Peak TNF-alpha Values as Categorized by Race and Gender
Time Frame: Baseline (-15 min, -5 min), and 1, 2, 4, 6, 12, 18, and 24 hours post LPS
Population: This analysis population was categorized by race and gender as follows: European American (EA) male n=102, African American (AA) male n=41, EU female n=91, and AA female n=60. Results include measurements at baseline and peak levels of Tumor Necrosis Factor- alpha (TNF-alpha).
Measure: Median (Inter-Quartile Range); unit: pg/ml
Groups:
- Niacin/Endotoxin: Niacin/Endotoxin: Subjects receive a one-time 1000mg dose of immediate release Niacin (Niacor pills), a one-time 1000mg dose of extended release Niacin (Niaspan pill) and one-time 1ng/kg injection of endotoxin (LPS).
Arm/Group | Niacin/Endotoxin
Number analyzed (Participants) | 294
pg/ml
  Baseline TNF-alpha in EA males (n=102) | 1.08 [0.9 to 1.51]
  Peak TNF-alpha in EA males (n=102) | 43.48 [23.38 to 67.08]
  Baseline TNF-alpha in AA males (n=41) | 1.03 [0.73 to 1.37]
  Peak TNF-alpha in AA males (n=41) | 37.28 [17.78 to 51.64]
  Baseline TNF-alpha in EA females (n=91) | 1.06 [0.82 to 1.45]
  Peak TNF-alpha in EA females (n=91) | 43.23 [17.32 to 83.2]
  Baseline TNF-alpha in AA females (n=60) | 1.13 [0.8 to 1.71]
  Peak TNF-alpha in AA females (n=60) | 34.01 [19.1 to 58.06]

2. Secondary Outcome: Baseline and Peak C-Reactive Protein (CRP) Values as Categorized by Race and Gender
Time Frame: Baseline ( -15 min, -5 min), and 1, 2, 4, 6, 12, 18, and 24 hours post LPS
Population: This analysis population was categorized by race and gender as follows: European American (EA) male n=102, African American (AA) male n=41, EU female n=91, and AA female n=60. Results include measurements at baseline and peak levels of C-Reactive Protein (CRP).
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Niacin/Endotoxin
Number analyzed (Participants) | 294
mg/L
  Baseline CRP in EA males | 0.34 [0.17 to 0.8]
  Peak CRP in EA males | 17.8 [11.23 to 24.23]
  Baseline CRP in AA males | 0.54 [0.34 to 1.19]
  Peak CRP in AA males | 14.25 [9.97 to 21.05]
  Baseline CRP in EA females | 0.62 [0.33 to 1.73]
  Peak CRP in EA females | 15.9 [9.88 to 21.9]
  Baseline CRP in AA females | 0.71 [0.21 to 1.92]
  Peak CRP in AA females | 10.8 [8.18 to 16.1]

ADVERSE EVENTS:
Time Frame: AE data collected for approximately 3.5 years, during the course of all study visits
Arm/Group | Niacin and Endotoxin
Serious Adverse Events (participants affected / at risk) | 0/400
Other Adverse Events (participants affected / at risk) | 86/400
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niacin and Endotoxin (N=400)
Headache (Nervous system disorders) | 13 (13)
Vomitting (Gastrointestinal disorders) | 28 (28)
Diarrhea (Gastrointestinal disorders) | 12 (12)
>2g drop in Hgb or <10 g/dL (Blood and lymphatic system disorders) | 18 (18) — > 2g drop in Hgb from baseline or <10 g/dL Hgb at discharge
Lightheadedness (Cardiac disorders) | 15 (15) — subject reported lightheadedness or dizziness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes